CLINICAL TRIAL: NCT00000806
Title: A Phase I Randomized Dose/Formulation Comparison Study of SC-52151
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: ACTG 282
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1995-02

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; HIV Protease Inhibitors
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex

INTERVENTIONS:
Drug: Telinavir

SUMMARY:
PRIMARY: To evaluate the safety, tolerability, pharmacokinetics, and ethanol exposure of two dose regimens and formulations of SC-52151.

SECONDARY: To evaluate the preliminary anti-HIV activity of these treatment regimens and the relationship between day 14 plasma concentrations of SC-52151 and immunological and virological markers and toxicity.

Since viral isolates with decreased susceptibility to the protease inhibitor SC-52151 occur in vitro after multiple passages, and since prolonged post infectious effects occur in vitro, comparison of two formulations, an elixir and a self-emulsifying drug delivery system (SEDDS), is needed to determine the appropriate dose formulation for Phase II studies.

DETAILED DESCRIPTION:
Since viral isolates with decreased susceptibility to the protease inhibitor SC-52151 occur in vitro after multiple passages, and since prolonged post infectious effects occur in vitro, comparison of two formulations, an elixir and a self-emulsifying drug delivery system (SEDDS), is needed to determine the appropriate dose formulation for Phase II studies.

Patients are randomized to four treatment arms to receive SC-52151 elixir or SEDDS formulation at 1 of 2 doses for 2 weeks, with follow-up for 14 days.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required for patients with CD4 count <= 200 cells/mm3:

* PCP prophylaxis using TMP/SMX or aerosolized pentamidine.

Allowed:

* Topical antifungal agents.
* Up to 1000 mg/day acyclovir as maintenance therapy for herpes simplex virus.
* Antibiotics for bacterial infections.
* Antipyretics, analgesics, nonsteroidal anti-inflammatory agents, antiemetics, and methadone for symptomatic treatment.

Patients must have:

* HIV infection.
* CD4 count 150 - 500 cells/mm3.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Unable to tolerate the standard diet required for the study.
* Unable to give informed consent.

Concurrent Medication:

Excluded:

* Antiretrovirals and biologic response modifiers (including HIV vaccines).
* Maintenance with ketoconazole, fluconazole, itraconazole, ganciclovir, foscarnet, pyrimethamine, sulfadiazine, clindamycin, azithromycin, isoniazid, rifampin, rifabutin, ethambutol, pyrazinamide, clofazimine, or clarithromycin.
* Prophylaxis for Mycobacterial infection or fungal infections other than Candidiasis.
* Allopurinol.
* Omeprazole.
* Astemizole.
* Terfenadine.
* Loratadine.
* Psychotropics.
* Phenylbutazone.
* Barbiturates.
* Benzodiazepines.
* Monoamine oxidase inhibitors.
* H-2 blockers.
* Anticonvulsants.
* Coumadin anticoagulants.
* Oral contraceptives.
* Antiarrhythmics.
* Diltiazem.
* Metronidazole.
* Erythromycin.
* Chloramphenicol.
* Fluoroquinolones.
* Disulfiram.
* Erythropoietin.
* G-CSF or GM-CSF.
* Systemic corticosteroids.
* Alcohol, including alcohol-containing medications.

Patients with the following prior conditions are excluded:

* Unexplained temperature >= 38.5 C for any 7 days within the 30 days prior to study entry.
* Chronic diarrhea (>= three stools per day) for any 15 days within the 30 days prior to study entry.
* Malignancy other than basal or squamous cell carcinoma of the skin, cervical intraepithelial neoplasia, and minimal Kaposi's sarcoma.

Prior Medication:

Excluded at any time:

* Prior HIV protease inhibitor.

Excluded within 30 days prior to study entry:

* Investigational drugs.
* Recombinant erythropoietin.
* G-CSF or GM-CSF.
* Interferon or interleukin.
* Any HIV-1 vaccine.

Excluded within 14 days prior to study entry:

* Antiretrovirals.
* Acute therapy for any opportunistic or other serious infection.
* Therapy for malignancy.
* Maintenance with ketoconazole, fluconazole, itraconazole, ganciclovir, foscarnet, pyrimethamine, sulfadiazine, clindamycin, azithromycin, isoniazid, rifampin, rifabutin, ethambutol, pyrazinamide, clofazimine, or clarithromycin.
* Prophylaxis for Mycobacterial infection or fungal infections other than Candidiasis.

Excluded within 7 days prior to study entry:

* Allopurinol.
* Omeprazole.
* Astemizole.
* Terfenadine.
* Loratadine.
* Psychotropics.
* Phenylbutazone.
* Barbiturates.
* Benzodiazepines.
* Monoamine oxidase inhibitors.
* H-2 blockers.
* Anticonvulsants.
* Coumadin anticoagulants.
* Oral contraceptives.
* Antiarrhythmics.
* Diltiazem.
* Metronidazole.
* Erythromycin.
* Chloramphenicol.
* Fluoroquinolones.
* Disulfiram.

Risk Behavior: Excluded:

* History of substance or alcohol abuse.
* Ingestion of more than 50 g alcohol daily within 6 months prior to study entry.
* Recovered alcoholic.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48

CONTACTS AND LOCATIONS:
Overall Officials: Fischl MA, Study Chair; Richman DD, Study Chair; Flexner C, Study Chair; Para MF, Study Chair
Locations (4):
- United States (4):
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Univ of Miami School of Medicine, Miami, Florida
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Ohio State Univ Hosp Clinic, Columbus, Ohio

REFERENCES:
- [Background] Fischl MA, Richman DD, Flexner C, Meehan P, Para MF, Haubrich R, Cook J, Wood K, Karim A. Phase I study of two formulations and dose schedules of SC- 521151, A protease inhibitor. Natl Conf Hum Retroviruses Relat Infect (2nd). 1995 Jan 29-Feb 2:88